CLINICAL TRIAL: NCT04364321
Title: The Efficacy of A Single Dose Clonazepam Compared With the Intermittent Diazepam to Prevent Recurrent Febrile Seizures in Queen Sirikit National Institute of Child Health
Brief Title: Single Dose of Clonazepam Versus Intermiittent Diazepam for Febrile Seizures Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Sirikit National Institute of Child Health (Other Government)
Responsible Party: Principal Investigator, Kullasate Sakpichaisakul, Director of Pediatric Neurology, Queen Sirikit National Institute of Child Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: QSNICH63-017
Record Dates: First submitted 2020-04-05; First posted 2020-04-28 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Recurrent Febrile Convulsion
Keywords: recurrent febrile convulsions; Clonazepam; prophylaxis
MeSH Terms: conditions — Seizures, Febrile | interventions — Clonazepam; Diazepam

STUDY DESIGN:
Intervention Model Description: A pragmatic parallel group randomized trial comparing single dose clonazepam with intermittent oral diazepam for prevention recurrent febrile seizures
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose Clonazepam (Experimental): Clonazepam(0.5 mg/tablet) 0.02 mg/kg orally once at the time of fever present. (body temperature more than 38 degree Celsius)
  Interventions: Drug: Clonazepam 0.5 MG
- Intermittent oral diazepam (Active Comparator): Diazepam 0.3 mg/kg every 8 hours for 3 doses. (24 hr) start at the time of body temperature more than 38 degree Celsius.
  Interventions: Drug: Diazepam Tablets

INTERVENTIONS:
Drug: Clonazepam 0.5 MG — Clonazepam 0.02 mg/kg only one dose
  Other Names: Rivotril; Povanil
  Arms: Single dose Clonazepam
Drug: Diazepam Tablets — Diazepam 0.3 mg/kg every 8 hours for 3 doses. (24 hr)
  Arms: Intermittent oral diazepam

SUMMARY:
To study the efficacy and safety of single dose clonazepam compared with intermittent oral diazepam for prevention of recurrent febrile seizures in children who had three or more febrile seizures.

DETAILED DESCRIPTION:
Febrile seizures are the most common type of seizures disorder of young children. The risk of recurrences are 33 percent overall, half of them had at least one recurrent seizure (the 3rd febrile seizures). After that the recurrent rate is 50-100 percent depend on their risk factors. A few studies found that multiple recurrent febrile seizures might associated with language developmental delayed, poor speed performance quotient, Attention deficit hyperactivity disorders. Moreover, seizures are upsetting both parents and children. During the febrile illness, the intermittent diazepam, continuous phenobarbital and valproate are effective for prevention of the recurrences. Because of the benign nature of a simple febrile seizures, the risks of side effects generally outweigh the benefits. However, there is no clinical guidelines for prevention of recurrent febrile seizures in the children who experienced multiple occurrences. The better prophylactic drug; safe, effective and easy to use, for prevention of recurrent febrile seizures in children with multiple recurrences might be needed. Clonazepam, the long half-life benzodiazepine, is commonly used for treatment of epilepsy may be effective in preventing recurrent febrile seizures. This study, a single-blind, randomized clinical trial, single dose clonazepam at the time of fever present compared with oral diazepam during the fever to prevent the recurrent febrile seizures.

ELIGIBILITY:
Inclusion Criteria:

* age 6-60 months at date of enrollment
* 3 or more episodes of clinically diagnosed febrile seizures

Exclusion Criteria:

* history of afebrile seizures or any history suggested the epilepsy
* history of previous brain insults; CNS infection, birth trauma, traumatic brain injury.
* delayed developmental milestones
* abnormal neurological examinations
* currently treatment by continous antiepileptic drug(s)
* A contraindication to Clonazepam, Diazepam such as drug hypersensitivity, liver disease.
* Predictable lack of available of follow up.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Recurrent rate of febrile seizures | the assessment will be done at 12 months after enrollment
  Rate of seizure occurs when the children have febrile illnesses (at the onset of fever until fever gone). The seizures will be reported by their parents/caregivers. (via the seizure record form and the interview.) Statistic analysis: Cumulative incidence (person-year). percent. Comparison between the two group by unpaired t test.

SECONDARY OUTCOMES:
Number of participants with adverse reaction of medications | 7 days
  The adverse reactions will be recorded by their caregivers in the record form for 7 days since patients taking the medication (clonapam or diazepam).
  The adverse reactions are drowsiness, ataxia, irritability, drooling, insomnia and rashes.
  Statistic analysis: cumulative incidence (person-year), Comparison between the two group by unpaired t test.
Associated factors: Sex | at the enrollment.
  To evaluate the associated factors of multiple recurrent febrile seizures.
  The data will be collected in the record form by the primary investigator at the enrollment.
  Statistic analysis: comparison between group by chi square
Associated factors: age at first febrile seizure | at the enrollment
  To evaluate the associated factors of multiple recurrent febrile seizures.
  The data will be collected in the record form by interviewing the caregivers to recall the information.
  Statistic analysis: comparison between group by unpaired t test
Associated factors: the lowest temperature that cause seizure | at the enrollment.
  To evaluate the associated factors of multiple recurrent febrile seizures.
  The data will be collected in the record form by interviewing the caregivers to recall the information.
  Statistic analysis: comparison between group by unpaired t test
Number of participants with febrile convulsions in parents or siblings | at the enrollment.
  To evaluate the associated factors of multiple recurrent febrile seizures.
  The data will be collected in the record form by interviewing the caregivers.
  Statistic analysis: comparison between group by chi square
Number of participants with epilepsy in parents or siblings | at the enrollment.
  To evaluate the associated factors of multiple recurrent febrile seizures.
  The data will be collected in the record form by interviewing the caregivers.
  Statistic analysis: comparison between group by chi square
Number of participants with type of febrile seizures (simple or complex) | at the enrollment.
  To evaluate the associated factors of multiple recurrent febrile seizures.
  Type of febrile seizure
  1. simple: seizure duration less than 15 min, generalized seizures, one seizure in 24 hours
  2. complex:15 minutes or more and/or focal seizures and/or 2 or more seizures in 24 hours
  The data will be collected in the record form by interviewing the caregivers.
  Statistic analysis: comparison between group by chi square
Number of participants with delayed developmental milestones | at the enrollment.
  The data will be collected by the developmental screening tools; Age and Stages Questionaires, third edition reported by the caregivers. Scoring will be done by neurology pediatrician at the enrollment.
  Age and Stages Questionaires(third editon) are divided in 5 areas; communication, gross motor, fine motor, problem solving, personal-social, each area has 6 questions. Scores for each area are between 0 to 60. The Cutoff points are different in each area. If the score is above the cutoff, the children development appears normal for age.
  (The cutoff for communication is 29.65, Gross motor is 22.25, fine motor is 25.14, problem solving is 27.72 and personal-social is 25.34)
  Statistic analysis: comparison between group by unpaired t test

CONTACTS AND LOCATIONS:
Overall Officials: Jinjutha Nithiuthai, MD, Principal Investigator — Queen Sirikit National Institute of Child Health
Locations (1):
- Queen Sirikit National Institute of Child Health, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available due to the confidentiality.

REFERENCES:
- [Background] Berg AT, Shinnar S, Darefsky AS, Holford TR, Shapiro ED, Salomon ME, Crain EF, Hauser AW. Predictors of recurrent febrile seizures. A prospective cohort study. Arch Pediatr Adolesc Med. 1997 Apr;151(4):371-8. doi: 10.1001/archpedi.1997.02170410045006. PMID 9111436
- [Background] Berg AT, Shinnar S, Hauser WA, Leventhal JM. Predictors of recurrent febrile seizures: a metaanalytic review. J Pediatr. 1990 Mar;116(3):329-37. doi: 10.1016/s0022-3476(05)82816-1. PMID 2137875
- [Background] Kolfen W, Pehle K, Konig S. Is the long-term outcome of children following febrile convulsions favorable? Dev Med Child Neurol. 1998 Oct;40(10):667-71. doi: 10.1111/j.1469-8749.1998.tb12326.x. PMID 9851235
- [Background] Visser AM, Jaddoe VW, Ghassabian A, Schenk JJ, Verhulst FC, Hofman A, Tiemeier H, Moll HA, Arts WF. Febrile seizures and behavioural and cognitive outcomes in preschool children: the Generation R study. Dev Med Child Neurol. 2012 Nov;54(11):1006-11. doi: 10.1111/j.1469-8749.2012.04405.x. Epub 2012 Sep 3. PMID 22937894
- [Background] Bertelsen EN, Larsen JT, Petersen L, Christensen J, Dalsgaard S. Childhood Epilepsy, Febrile Seizures, and Subsequent Risk of ADHD. Pediatrics. 2016 Aug;138(2):e20154654. doi: 10.1542/peds.2015-4654. Epub 2016 Jul 13. PMID 27412639
- [Background] Billstedt E, Nilsson G, Leffler L, Carlsson L, Olsson I, Fernell E, Gillberg C. Cognitive functioning in a representative cohort of preschool children with febrile seizures. Acta Paediatr. 2020 May;109(5):989-994. doi: 10.1111/apa.15059. Epub 2019 Nov 10. PMID 31618476
- [Result] Rosman NP, Colton T, Labazzo J, Gilbert PL, Gardella NB, Kaye EM, Van Bennekom C, Winter MR. A controlled trial of diazepam administered during febrile illnesses to prevent recurrence of febrile seizures. N Engl J Med. 1993 Jul 8;329(2):79-84. doi: 10.1056/NEJM199307083290202. PMID 8510706
- [Result] Knudsen FU. Recurrence risk after first febrile seizure and effect of short term diazepam prophylaxis. Arch Dis Child. 1985 Nov;60(11):1045-9. doi: 10.1136/adc.60.11.1045. PMID 3907504
- [Result] Capovilla G, Mastrangelo M, Romeo A, Vigevano F. Recommendations for the management of "febrile seizures": Ad Hoc Task Force of LICE Guidelines Commission. Epilepsia. 2009 Jan;50 Suppl 1:2-6. doi: 10.1111/j.1528-1167.2008.01963.x. PMID 19125841
- [Result] Offringa M, Newton R, Cozijnsen MA, Nevitt SJ. Prophylactic drug management for febrile seizures in children. Cochrane Database Syst Rev. 2017 Feb 22;2(2):CD003031. doi: 10.1002/14651858.CD003031.pub3. PMID 28225210